CLINICAL TRIAL: NCT02509390
Title: Hyperfibrinogenemia Within the First Days After Major Trauma : Kinetic, Functionality, Impact of Fibrinogen Replacement Therapy and Trauma, Thrombosis Risk
Brief Title: Hyperfibrinogenemia After Major Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9239
Record Dates: First submitted 2013-12-10; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Major Trauma
Keywords: Fibrinogen level; Hyperfibrinogenemia; Trauma; Thrombosis risk
MeSH Terms: conditions — Wounds and Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Severe trauma patients (Experimental): All severe trauma patients (ISS>15) admitted in our trauma center Blood samples (additional blood tubing)
  Interventions: Procedure: Blood samples

INTERVENTIONS:
Procedure: Blood samples — Investigators analyze hematological parameters with blood sampled daily in severe trauma patients

SUMMARY:
Assessment of the evolution of fibrinogen plasma level within the first ten days after major trauma in order to determine prevalence of hyperfibrinogenemia (Fg > 4 g/L) and its time to onset.

DETAILED DESCRIPTION:
In this study, investigators daily investigate fibrinogen plasma levels and fibrinogen antigen in severe trauma patients (Injury severity score > 15) within the first ten days. Investigators then modelize hyperfibrinogenemia profiles according to severity of injuries and physiopathologic mechanisms. Finally, investigators determine predisposing risk factors to develop hyperfibrinogenemia and assess the impact of fibrinogen replacement therapy in initial phase of management of major trauma.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old.
* Polytrauma with ISS Score > 15
* Hospitalized patients in reanimation unit < 4h after trauma
* Informed consent

Exclusion Criteria:

* Patients in another study
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
daily fibrinogen level >4 g/L | 10 days
  the occurrence and delay of fibrinogen level > 4 g/L after major trauma

SECONDARY OUTCOMES:
assessing predisposing risk factors of hyperfibrinogenemia (> 4 g/l) | 10 days
  Initial chock status severity, vascular filling, initial acidose, hypothermia, trauma severity (ISS scores, Sequential Organ Failure Assessment (SOFA), IGS2), numbers and sites of lesions (AIS scores), severity of initial failure of fibrinogene, administration of fibrinogene at initial hemorrhagic phase…
plasmatic fibrinogen level evolution | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Pauline PD DERAS, MD, Principal Investigator — Regional Trauma Center, Department of Anesthesiology and critical care, Lapeyronie University Hospital, Montpellier
Locations (1):
- Department of Anesthesiology and critical care, Lapeyronie University Hospital, Montpellier, France